CLINICAL TRIAL: NCT02616081
Title: Patient Reported Outcomes for Bladder Management Strategies in Spinal Cord Injury
Acronym: NBRG-PCORI
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Minnesota (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Jeremy Myers, Associate Professor - School of Medicine, University of Utah
Other Study IDs: 82971
Record Dates: First submitted 2015-11-13; First posted 2015-11-26 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Neurogenic Bladder; Spinal Cord Injuries; Quality of Life; Incontinence
Keywords: Urinary Bladder; Neurogenic; Quality of Life; Spinal cord injury; incontinence; Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries | interventions — Intermittent Urethral Catheterization; Catheters, Indwelling; Surgical Procedures, Operative; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Clean Intermittent Catheterization: Participants performing intermittent catheterization of their bladder, having not had augmentation cystoplasty or creation of a catheterizable channel
  Interventions: Other: Clean Intermittent Catheterization
- Indwelling Catheter: Participants utilizing an Foley catheter or a suprapubic tube (cystostomy)
  Interventions: Other: Indwelling Catheter
- Surgery: Undergoing any of the following surgeries: augmentation cystoplasty with or without a catheterizable channel, creation of catheterizable channel alone, urinary diversion (conduit or continent catheterizable pouch)
  Interventions: Other: Surgery
- Voiding: Participants with volitional control, voiding into diapers or a condom catheter via crede, valsalva, or spontaneous leakage
  Interventions: Other: Voiding

INTERVENTIONS:
Other: Clean Intermittent Catheterization — Clean intermittent self catheterization is a standard of care.
  Groups: Clean Intermittent Catheterization
Other: Indwelling Catheter — Indwelling catheterization is a standard of care.
  Groups: Indwelling Catheter
Other: Surgery — Bladder surgery is a standard of care.
  Groups: Surgery
Other: Voiding — Voiding spontaneously is a standard of care.
  Groups: Voiding

SUMMARY:
The investigators goal is to create a better understanding of patient reported outcomes for bladder management strategies (clean intermittent catheterization (CIC), indwelling catheter (IDC) and bladder surgery.

DETAILED DESCRIPTION:
Our study is a longitudinal observational study between bladder management strategies, comparing outcomes measured by patient reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants with acquired spinal cord injury
* Participants with neurogenic bladder
* Participants must be undergoing or starting at least one of the following bladder management treatments at the time of enrollment. a) Clean intermittent catheterization (CIC) b) Have an indwelling catheter (IDC) c) Spontaneous voiding, and d) Have undergone bladder surgery
* Age 18 or older
* Willingness and ability to comply with study engagement
* Able to provide consent

Exclusion Criteria:

* Degenerative spinal cord issues, such as multiple sclerosis, neuromuscular dysfunction
* Congenital spinal cord issues, such as spina bifida, myelomeningocele, or cerebral palsy
* Participants that belong to a vulnerable population (pregnant, prisoners, mentally handicapped, etc)
* Participants less than 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with neurogenic bladder with urinary issues and currently being managed by one/ any of various bladder management treatments (clean intermittent catheterization, indwelling catheter, voiding or bladder surgery).
Sampling Method: Non-Probability Sample
Enrollment: 1479 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Neurogenic Bladder Symptom Score (NBSS): comparing change in: CIC, IDC, Voiding, and Surgery | Baseline and 1 year longitudinal follow up
  The NBSS quantifies bladder symptoms
The Spinal Cord Injury Quality of Life Measurement System Bladder Management Difficulties (SCI-QOL Difficulties): comparing change in: CIC, IDC, Voiding, and Surgery | Baseline and 1 year longitudinal follow up
  The SCI-QoL Difficulties assesses feelings and psychosocial impact of bladder symptoms
The Spinal Cord Injury Quality of Life Measurement System Bladder Complications (SCI-QOL Complications): comparing change in: CIC, IDC, Voiding, and Surgery | Baseline and 1 year longitudinal follow up
  The SCI-QoL Complications assesses degree of bladder complications their psychosocial impact

SECONDARY OUTCOMES:
NBSS Incontinence subdomain | Baseline and 1 year longitudinal follow up
  The Incontinence subdomain measures degree of incontinence
NBSS Storage and Voiding subdomain | Baseline and 1 year longitudinal follow up
  The Storage and Voiding subdomain measures symptoms related to frequency and emptying of the bladder
NBSS Consequences subdomain | Baseline and 1 year longitudinal follow up
  The Consequences subdomain measures bladder related complications
NBSS QoL Satisfaction | Baseline and 1 year longitudinal follow up
  The final question of the NBSS assesses overall satisfaction with the urinary system

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy O Myers, MD, Principal Investigator — University of Utah School of Medicine - Urology
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patel DP, Lenherr SM, Stoffel JT, Elliott SP, Welk B, Presson AP, Jha A, Rosenbluth J, Myers JB; Neurogenic Bladder Research Group. Study protocol: patient reported outcomes for bladder management strategies in spinal cord injury. BMC Urol. 2017 Oct 10;17(1):95. doi: 10.1186/s12894-017-0286-3. PMID 29017505
- [Derived] Crescenze IM, Lenherr SM, Myers JB, Elliott SP, Welk B, O'Dell D, Stoffel JT. Self-Reported Urological Hospitalizations or Emergency Room Visits in a Contemporary Spinal Cord Injury Cohort. J Urol. 2021 Feb;205(2):477-482. doi: 10.1097/JU.0000000000001386. Epub 2020 Oct 9. PMID 33035138
- See also: Neurogenic Bladder Research Group — http://www.nbrg.org

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02616081/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT02616081/ICF_001.pdf